CLINICAL TRIAL: NCT03028701
Title: Assessment of Bronchodilator Efficacy of Formoterol/Budesonide 12/400 mcg Via Discair in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Assessment of Bronchodilator Efficacy of Formoterol/Budesonide 12/400 mcg Via Discair in COPD
Acronym: COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-20.13
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2017-01

CONDITIONS: Copd
Keywords: Formoterol; Budesonide; Dry powder inhalation; Discair; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Formoterol/Budesonide 12/400 mcg Discair (Experimental): Formoterol/Budesonide 12/400 mcg Inhalation Powder (1 puff) once daily via Discair®
  Interventions: Drug: Formoterol/Budesonide 12/400 mcg Discair

INTERVENTIONS:
Drug: Formoterol/Budesonide 12/400 mcg Discair — Formoterol/Budesonide 12/400 mcg Inhalation Powder (1 puff) once daily via Discair®
  Other Names: Forpack Discair® Inhalation Powder 12/400 mcg.

SUMMARY:
The overall objective is to asses the bronchodilator effect of single dose of Formoterol/Budesonide 12/400 mcg fixed combination delivered via Discair® in patients with COPD.

Spirometric measurements (FEV1, FVC) will be performed for a period of 12 h at 12 different times: pretreatment (prior to the first dose) and posttreatment (15. min, 30. min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr ve 12 hr).

DETAILED DESCRIPTION:
The overall objective is to asses the bronchodilator effect of single dose of Formoterol/Budesonide 12/400 mcg fixed dose combination delivered via Discair® in patients with COPD.

Patients will be assigned to receive single dose of Formoterol/Budesonide 12/400 mcg fixed dose combination delivered via Discair® (test product, n = 33). Patients will be evaluated at 4 consecutive visits: baseline (enrollment), screening, treatment, and end of treatment (24h after treatment).

For newly diagnosed and formerly diagnosed patients who are not on COPD medication, the screening visit will be performed on the day of enrollment. For formerly diagnosed patients receiving COPD treatment, the day of the screening visit will be based on the completion of a run-in period, with the length determined by the specific medication. During the run-in period, salbutamol (100 μg inhaler) will be prescribed as a rescue medication.

Spirometric measurements (FEV1, FVC) will be performed for a period of 12 h at 12 different times: pretreatment (prior to the first dose) and posttreatment (15. min, 30. min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr ve 12 hr).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years with newly or formerly diagnosed moderate to severe COPD (Patients with postbronchodilator FEV1/FVC ratio <0.70, and FEV1 <80% of predicted normal. Patients have chronic cough or chronic productive cough with breathlessness even walking slowly along flat ground.) Current smokers or exsmokers with a smoking history of at least 10 pack-years
* Patients who have no exacerbation within last 4 weeks
* Females patients with childbearing potential using effective birth control method
* Patients who has a capability of communicate with investigator
* Patients who accept to comply with the requirements of the protocol
* Patients who signed written informed consent prior to participation

Exclusion Criteria:

* Patients who have history of hypersensitivity to drugs contains long-acting beta2-agonist or corticosteroids
* Patients who have abnormal blood glucose level ((≥140 mg/dl)
* Patients who have unregulated diabetes mellitus
* Patients who have a serum potassium level of ≤3.5 mEq/L or >5.5mEq/L
* Patients who have asthma
* Patients who have a history of myocardial infarction, severe hearth failure, acute ischemic coroner disease or severe cardiac arrhythmia requiring treatment within least 6 weeks
* Patients who have lung cancer
* Patients vaccinated with live attenuated vaccines within 2 weeks prior to screening visit or during run-in period.
* Patients who had COPD exacerbation or lower respiratory track infections that required antibiotic, oral or parenteral corticosteroid treatment within 4 weeks prior to screening visit or during run-in period.
* Women who are pregnant or nursing
* History of allergic rhinitis or atopy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Mean max improvement (ml) from baseline in FEV1 over a period of 12 h. | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
The time to onset of max improvement from baseline in FEV1. | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.

SECONDARY OUTCOMES:
Mean absolute change (ml) from baseline in FEV1 over a period of 12 h (over spirometric measurement period). | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
Mean absolute change (ml) from baseline in FVC over a period of 12 h (over spirometric measurement period). | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
Mean % change from baseline in FEV1 over a period of 12 h (over spirometric measurement period). | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
Mean % change from baseline in FVC over a period of 12 h (over spirometric measurement period). | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
FEV1 (AUC0-12) response | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
FVC (AUC0-12) response | Pretreatment (prior to the first dose of study medication) and posttreatment (Day 1)
  Spirometric measurements will be made at prior to the first dose of study medication and and posttreatment at 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 8 hr, 10 hr and 12 hr.
Evaluation of safety | Predose and up to 12 hours postdose
  (Physical examination, numbers of adverse reactions and abnormal laboratory values related

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Yıldız, Assoc. Prof., Principal Investigator — Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital Istanbul, Turkey, 34020
Locations (1):
- Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildiz P, Bayraktaroglu M, Gorgun D, Yuksel K. Bronchodilator Efficacy of a Single-Dose 12/400-microg Formoterol/Budesonide Combination as a Dry Powder for Inhalation Delivered by Discair(R) in Adult Patients with Moderate-to-Severe Stable COPD: Open-Label, Single-Arm, Phase IV Trial. Clin Drug Investig. 2019 Oct;39(10):991-1001. doi: 10.1007/s40261-019-00828-y. PMID 31332649